CLINICAL TRIAL: NCT02626637
Title: KAM: Kids Are Moving; An Exercise Program for Children With Cancer
Brief Title: KAM: Kids Are Moving
Acronym: KAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1412M57161
Record Dates: First submitted 2015-11-25; First posted 2015-12-10 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Children With Cancer; Fatigue; Physical Activity
Keywords: children with cancer; fatigue; physical activity
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical activity coaching (Experimental): Children and adolescents will receive the study intervention, which includes exercise coaching and prescription, that is be incorporated into the standard care they receive from the nurse practitioners during their outpatient visits.
  Interventions: Other: Physical activity coaching

INTERVENTIONS:
Other: Physical activity coaching — Children and adolescents will receive the study intervention, which includes exercise coaching and prescription, that is be incorporated into the standard care they receive from the nurse practitioners during their outpatient visits.

SUMMARY:
During cancer treatment children are less active than their health peers. This inactivity persists into survivorship and can negatively affect health and quality of life. Physical activity may also improve fatigue, a prevalent and distressing symptom during treatment. Improving health behaviors during treatment can have lifelong benefits for cancer survivors. In this study, the effectiveness of the "Kids are Moving" exercise program will be evaluated. The exercise program will follow program guidelines set up by the American College of Sports Medicine and will be adapted for children with cancer. Children ages 6 to 18 years, who are receiving chemotherapy, and their parents, will be coached on how to increase their physical activity and will receive an exercise prescription. This will occur as part of the standard care they receive from the nurse practitioners during the first six months of their outpatient visits. Investigators want to find out if children in the Kids are Moving program are more active and have less fatigue. Activity will be measured through patient questionnaires about activity and fatigue, and by wearing the FitBit activity tracker and an actigraph. Outcomes will be compared to measurements collected from children who received usual care before the exercise program started.

Physical activity is a vital for improving health and quality of life and for providing energy for engaging in positive life experiences as children move along the developmental continuum to a long and healthy future. Outcomes of the study will provide a foundation for larger multi-site clinical trials.

DETAILED DESCRIPTION:
During cancer treatment children are significantly less active than their healthy peers. This inactivity persists into survivorship, negatively influencing their health and quality of life. Physical activity may also improve fatigue, a near-universal and distressing symptom during treatment. Improving health behaviors during treatment can have lifelong benefit.

The goal of this study is to evaluate the effectiveness of the Kids are Moving exercise program that is delivered by nurse practitioners (NP's) during outpatient care provided to a specific population of children. The study will be conducted at two pediatric cancer treatment sites and will translate the American College of Sports Medicine's program, Exercise is Medicine into practice. In this quasi-experimental design, children will receive the study intervention, which includes exercise coaching and prescription, that is be incorporated into the standard care they receive from the nurse practitioners during their outpatient visits. Outcomes will be compared to historical control measurements of children who received usual care. Study aims are to:

1. To compare measurements of activity levels of children receiving exercise coaching over the first 6 months of cancer treatment as measured by self-report and the FitBit Flex tracker
2. To compare activity levels of children receiving exercise coaching during cancer treatment as measured by self-report and the FitBit Flex tracker, to activity levels of children in the historical control group receiving usual care during cancer treatment.
3. To evaluate the influence of activity levels on fatigue experience by children receiving cancer treatment

Children ages 6 to 18, and their parents, will be invited to participate in study measurements which will be completed at the 2nd, 4th, and 6th months of cancer treatment. Patients will be included if recently diagnosed with cancer (excluding bone tumors and bone metastasis), and ambulatory. Validated self-report instruments will be used to measure activity and fatigue. Additionally, the FitBit Flex tracker, a device that measures steps/day and motion in three dimensions and an actigraph, will be worn by subjects over a 3 day period for each measurement point.

Physical activity is a vital intervention for improving health and quality of life and for providing energy for engaging in positive life experiences that advance children along the developmental continuum to a long and healthy future. Outcomes of the study will provide a foundation for larger multi-site clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 6 and 18 with any cancer diagnosis except for bone tumors or have bone metastasis
2. have received cancer treatment that includes chemotherapy for at least 2 months, have outpatient visits at least once a month, and are ambulatory
3. speak English
4. are able to give assent according to institutional guidelines
5. have parental consent to participate.

Exclusion Criteria:

1. Not meeting inclusion criteria

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Physical activity measured by FitBit Flex | Change from Baseline, at 2 month, at 4, months, at 6 months

SECONDARY OUTCOMES:
Self-report of fatigue | Change from Baseline, at 2 month, at 4, months, at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Casey C Hooke, PhD, APRN, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - Children's Minnesota, Minneapolis, Minnesota
  - University of Minnesota Masonic Childrens, Minneapolis, Minnesota